CLINICAL TRIAL: NCT04298957
Title: See and Treat in an Outpatient Setting in Women Above 45 Years With Cervical Dysplasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 172230
Record Dates: First submitted 2020-02-03; First posted 2020-03-06 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2021-04

CONDITIONS: Cervical Dysplasia; Cervical Lesion; Cervix Disease
Keywords: Cone biopsy; Colposcopy; See and treat
MeSH Terms: conditions — Uterine Cervical Dysplasia; Uterine Cervical Diseases | interventions — Conization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- See and treat (Other): Cone biopsi is offered to women age ≥ 45 years referred to Department of Obstetrics and Gynecology due to a positive cervical screening test and partly or invisible transformation zone.
  Interventions: Procedure: Cone biopsy

INTERVENTIONS:
Procedure: Cone biopsy — Cone biopsy if transformation Zone (TZ) 2 or TZ 3

SUMMARY:
The study will investigate if implementation of "see and treat" in the outpatient clinic can optimize the diagnosis, clinical follow-up and treatment of older women with positive cervical screening test.

DETAILED DESCRIPTION:
In Denmark, 370 women are diagnosed with cervical cancer every year and approximately 100 women die from the disease. Young women can be protected with the HPV vaccine, but it will take decades before the vaccine has an effect on older women. Women who are HPV positive have a risk of developing severe dysplasia of 25-55% within 10 years. Compared to younger women, older women are also more likely to be diagnosed with advanced-stage disease and their mortality is high. Due to retraction of the transformation zone into the cervical canal and atrophy of the mucosa the performance of colposcopy is low. Furthermore, the sensitivity of cytology decreases with age. This makes it very difficult to obtain sufficient biopsies and therefore postmenopausal women are often required to undergo colposcopy two to three times. Waiting for a final diagnosis and treatment not only has a large mental and practical impact on the women themselves, but it is also an economic burden for the health care system.

"See and treat" is a procedure that involves cervical cytology and HPV test, a colposcopy, cervical biopsies, and finally a loop electrosurgical excisional procedure by which the transformation zone is removed. This approach allows women to be diagnosed and treated in one visit.

In this project, the aim is to investigate if the implementation of "see and treat" in a gynecological outpatient clinic can optimize the diagnostics, clinical follow-up, and treatment of older women with abnormal cervical cytology or HPV-infection.

Participants Women aged ≥ 45 years with cervical dysplasia and/or a positive HPV test are referred from the general practitioner to the gynecological department.

Procedure At each inclusion site, the local project manager evaluates all the referred women for possible inclusion. Project information is sent either by e-mail or letter to eligible women. At the outpatient clinic, the eligible women will be informed about the project and asked to sign an informed consent form regarding their participation in the project.

If the eligible women agree to participate a physician in the outpatient clinic will obtain a cervical smear (i.e. cytology and Human Papillomavirus (HPV) test) and perform colposcopy and take four random biopsies. If the transformation zone (TZ) is partly visible or not visible a cone biopsy will be performed in local anesthesia (Citanest).

If the participant meet the exclusion criteria or declines to participate standard treatment will be offered (colposcopy and biopsies).

The included patients will be followed up with an HPV test after 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥ 45 years with a positive screening test (abnormal cytology and/or persistence HPV positive) who are referred to the Department of Obstetrics and Gynecology.
* Type 2 or 3 transformation zone (a partly or invisible transformation zone).

Exclusion Criteria:

* Type 1 transformation zone (fully visible)
* Current or previous diagnosis of cervical cancer.
* Pregnancy or pregnancy wish.
* Previously cone biopsy

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2019-03-13 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Cervical intraepithelial neoplasia ≥ grade 2 (CIN2+) lesion after referral with a positive cervical screening test | The histological diagnose from the Pathological Department will be available 8 weeks after inclusion.
  The prevalence of CIN2+ lesions in women ≥45 years included in the study
Concordance between cytology and histology | The histological diagnose from the Pathological Department will be available 8 weeks after inclusion.
  Concordance between cytology, biopsies and cone biopsy in the ability to detect CIN2+ changes
Clearance of HPV | This will be available 7 months after inclusion.
  Clearance rate of HPV after 6 months
Complication rate | Complication rate will be evaluated 6 months after inclusion.
  Complication rate of bleeding, infection and/or stenosis

CONTACTS AND LOCATIONS:
Overall Officials: Line W Gustafson, MD, Principal Investigator — Randers Regional Hospital and Aarhus University
Locations (3):
- Denmark (3):
  - Horsens Regional Hospital, Horsens, Jutland
  - Randers Regional Hospital, Randers, Jutland
  - Viborg Regional Hospital, Viborg, Jutland

IPD SHARING:
Plan to Share IPD: No
The dataset generated and analyzed in this study are not available for the public due to Danish legislation.

REFERENCES:
- [Derived] Binderup KO, Boers J, Gustafson LW, Andersen B, Petersen LK, Bor P, Gribnau J, Quint WGV, Van Den Munckhof H, Tranberg M, Hammer A. DNA-Methylation for Risk-Stratification of Women Without a Fully Visible Transformation Zone at Colposcopy: A Cross-Sectional Study. BJOG. 2025 Jul 14. doi: 10.1111/1471-0528.18288. Online ahead of print. PMID 40654017
- [Derived] Hammer A, Gustafson LW, Christensen PN, Brondum R, Andersen B, Andersen RH, Tranberg M. Implementation of p16/Ki67 dual stain cytology in a Danish routine screening laboratory: Importance of adequate training and experience. Cancer Med. 2020 Nov;9(21):8235-8242. doi: 10.1002/cam4.3399. Epub 2020 Sep 7. PMID 32894896